CLINICAL TRIAL: NCT04239417
Title: Effect of Preoperative Graduated Abdominal Exercises and Russian Current Stimulation on Muscle Strength Post Ventral Hernioplasty
Brief Title: Effect of Preoperative Abdominal Exercises and Russian Current on Muscle Strength Post Ventral Hernioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Ph. D Candidate., Assistant Lecturer, South Valley University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002036
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Muscle Strength
Keywords: ventral hernia; graduated abdominal exercises; isokinetic dynamometer.
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Sixty patients with ventral hernia, preoperatively, were randomly distributed into four equal groups: groups (A) & (B) & (C) ( three study groups ) and group (D) ( control group ).
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: groups (A) & (B) & (C) ( three study groups ) and group (D) ( control group )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The Study group A (Experimental): graduated abdominal strengthening exercises group
  Interventions: Other: Graduated abdominal strengthening exercises
- The Study group B (Experimental): Russian stimulation group
  Interventions: Device: The Russian current stimulation
- The Study group C (Experimental): combination group
  Interventions: Combination Product: Graduated abdominal strengthening exercises and the Russian current stimulation
- The Control group D (No Intervention): presume in normal activities of daily living.

INTERVENTIONS:
Other: Graduated abdominal strengthening exercises — 1. Exercise mat and inflatable Swiss ball
  2. Wall bar, wedges, elastic tubing
  Arms: The Study group A
Device: The Russian current stimulation — The Russian current is used for enhancing muscle; the muscular fiber by the electric stimulation.
  Arms: The Study group B
Combination Product: Graduated abdominal strengthening exercises and the Russian current stimulation — Combination between The Russian current and abdominal exercises
  Arms: The Study group C

SUMMARY:
The study was conducted to investigate the effect of preoperative graduated abdominal strengthening exercises and Russian stimulation on the abdominal muscles strength after ventral hernioplasty by using isokinetic dynamometer and Ultrasonography as methods of measurement.

DETAILED DESCRIPTION:
The study was conducted to investigate the effect of preoperative graduated abdominal strengthening exercises and Russian stimulation on the abdominal muscles strength after ventral hernioplasty by using isokinetic dynamometer and Ultrasonography as methods of measurement.

ELIGIBILITY:
Criteria of inclusion:

* The age is from 20 to 45 years.
* All patients want to optionally repair surgery.
* Ventral hernia is diagnosed on the basis of a surgeon evaluation.
* The study will include all patients.
* The informed consent of all the patients enrolled.

Criteria for exclusion:

* history of surgical interference for less than one year (abdominal surgery).
* Cirrhosis of the liver with ascites or without them.
* Deformity or contracture of the hip or spine.
* Obstruction of bowel, peritonitis or drilling.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Abdominal muscles peak torque | first or initial assessment at day 0.
  Peak torque is the single highest torque output of the joint produced by muscular contraction as the limb moves through the range of motion.
Abdominal muscles peak torque | second or preoperative assessment after 6 weeks of treatment.
  Peak torque is the single highest torque output of the joint produced by muscular contraction as the limb moves through the range of motion.
Abdominal muscles peak torque | third assessment at 2 months post-operative.
  Peak torque is the single highest torque output of the joint produced by muscular contraction as the limb moves through the range of motion.
Abdominal muscles peak torque | fourth assessment at 4 months post-operative.
  Peak torque is the single highest torque output of the joint produced by muscular contraction as the limb moves through the range of motion.
Abdominal muscles thickness | first or initial assessment at day 0.
  it is a method for muscle strength measurement as muscle strength is correlated to its cross section or diameter.
Abdominal muscles thickness | second or preoperative assessment after 6 weeks of treatment.
  it is a method for muscle strength measurement as muscle strength is correlated to its cross section or diameter.
Abdominal muscles thickness | third assessment at 2 months post-operative.
  it is a method for muscle strength measurement as muscle strength is correlated to its cross section or diameter.
Abdominal muscles thickness | fourth assessment at 4 months post-operative.
  it is a method for muscle strength measurement as muscle strength is correlated to its cross section or diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E. Ali, PhD student, Principal Investigator — South Valley University, Faculty of Physical Therapy
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward AR, Shkuratova N. Russian electrical stimulation: the early experiments. Phys Ther. 2002 Oct;82(10):1019-30. PMID 12350217
- [Background] Aguirre DA, Santosa AC, Casola G, Sirlin CB. Abdominal wall hernias: imaging features, complications, and diagnostic pitfalls at multi-detector row CT. Radiographics. 2005 Nov-Dec;25(6):1501-20. doi: 10.1148/rg.256055018. PMID 16284131
- [Background] Ahmed U, Ahmed R, Kamat S, Elkholy K. An ovary as unusual contents of an incarcerated umbilical hernia. Ann R Coll Surg Engl. 2014 Sep;96(6):e4-5. doi: 10.1308/003588414X13946184901443. PMID 25198958
- [Background] de Carvalho Froufe Andrade AC, Caserotti P, de Carvalho CM, de Azevedo Abade EA, da Eira Sampaio AJ. Reliability of Concentric, Eccentric and Isometric Knee Extension and Flexion when using the REV9000 Isokinetic Dynamometer. J Hum Kinet. 2013 Jul 5;37:47-53. doi: 10.2478/hukin-2013-0024. eCollection 2013. PMID 24146704
- [Background] Deeken CR, Lake SP. Mechanical properties of the abdominal wall and biomaterials utilized for hernia repair. J Mech Behav Biomed Mater. 2017 Oct;74:411-427. doi: 10.1016/j.jmbbm.2017.05.008. Epub 2017 May 6. PMID 28692907
- [Result] Young MJ, Gorlin AW, Modest VE, Quraishi SA. Clinical implications of the transversus abdominis plane block in adults. Anesthesiol Res Pract. 2012;2012:731645. doi: 10.1155/2012/731645. Epub 2012 Jan 19. PMID 22312327
- [Result] Howell B, Medina LE, Grill WM. Effects of frequency-dependent membrane capacitance on neural excitability. J Neural Eng. 2015 Oct;12(5):056015-56015. doi: 10.1088/1741-2560/12/5/056015. Epub 2015 Sep 8. PMID 26348707
- [Result] Wang HQ, Wei YY, Wu ZX, Luo ZJ. Impact of leg lengthening on viscoelastic properties of the deep fascia. BMC Musculoskelet Disord. 2009 Aug 21;10:105. doi: 10.1186/1471-2474-10-105. PMID 19698092
- [Result] Vinstrup J, Sundstrup E, Brandt M, Jakobsen MD, Calatayud J, Andersen LL. Core Muscle Activity, Exercise Preference, and Perceived Exertion during Core Exercise with Elastic Resistance versus Machine. Scientifica (Cairo). 2015;2015:403068. doi: 10.1155/2015/403068. Epub 2015 Oct 18. PMID 26557405
- [Result] van Bemmel AJ, van Marle AG, Schlejen PM, Schmitz RF. Handlebar hernia: a case report and literature review on traumatic abdominal wall hernia in children. Hernia. 2011 Aug;15(4):439-42. doi: 10.1007/s10029-010-0665-0. Epub 2010 May 1. PMID 20437188
- [Result] Aboodarda SJ, Page PA, Behm DG. Muscle activation comparisons between elastic and isoinertial resistance: A meta-analysis. Clin Biomech (Bristol). 2016 Nov;39:52-61. doi: 10.1016/j.clinbiomech.2016.09.008. Epub 2016 Sep 20. PMID 27681867
- [Result] Allen WM, Xu Z, Asman AJ, Poulose BK, Landman BA. Quantitative Anatomical Labeling of the Anterior Abdominal Wall. Proc SPIE Int Soc Opt Eng. 2013 Mar 28;8673:867312. doi: 10.1117/12.2007071. PMID 24478827
- [Result] Becker I, Woodley SJ, Stringer MD. The adult human pubic symphysis: a systematic review. J Anat. 2010 Nov;217(5):475-87. doi: 10.1111/j.1469-7580.2010.01300.x. Epub 2010 Sep 14. PMID 20840351
- [Result] Campanelli G, Pettinari D, Cavalli M, Avesani EC. Inguinal hernia recurrence: Classification and approach. J Minim Access Surg. 2006 Sep;2(3):147-50. doi: 10.4103/0972-9941.27728. PMID 21187986
- [Result] Dur AH, den Hartog D, Tuinebreijer WE, Kreis RW, Lange JF. Low recurrence rate of a two-layered closure repair for primary and recurrent midline incisional hernia without mesh. Hernia. 2009 Aug;13(4):421-6. doi: 10.1007/s10029-009-0487-0. Epub 2009 Mar 19. PMID 19296196
- [Result] Ellenbecker TS, Davies GJ. The application of isokinetics in testing and rehabilitation of the shoulder complex. J Athl Train. 2000 Jul;35(3):338-50. PMID 16558647
- [Result] Porcari JP, Miller J, Cornwell K, Foster C, Gibson M, McLean K, Kernozek T. The effects of neuromuscular electrical stimulation training on abdominal strength, endurance, and selected anthropometric measures. J Sports Sci Med. 2005 Mar 1;4(1):66-75. eCollection 2005 Mar 1. PMID 24431963

DOCUMENTS (1):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT04239417/Prot_001.pdf